CLINICAL TRIAL: NCT05364684
Title: The Impact of Ibutamoren on Nonalcoholic Fatty Liver Disease: A Pilot Study
Brief Title: The Impact of Ibutamoren on Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Laura Dichtel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P001057
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: NAFLD; Nonalcoholic Fatty Liver; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ibutamoren mesylate

STUDY DESIGN:
Intervention Model Description: Open-label study with historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label Treatment (Other): Open-label study of oral LUM-201 (ibutamoren mesylate) 25mg daily in otherwise healthy adults with BMI ≥25 kg/m2 and histologic or radiologic diagnosis of NAFLD.
  Interventions: Drug: LUM-201

INTERVENTIONS:
Drug: LUM-201 — LUM-201 (ibutamoren mesylate) is an oral growth hormone secretagogue.
  Other Names: Ibutamoren Mesylate

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD), fatty infiltration of the liver in the absence of alcohol use, is an increasingly recognized complication of obesity, with prevalence estimates of about 30% of individuals in the United States. A subset of these will develop progressive disease in the form of nonalcoholic steatohepatitis (NASH), which can progress to cirrhosis and liver failure. The investigators hypothesize that LUM-201 (Ibutamoren mesylate) will decrease intrahepatic lipid accumulation as quantified by proton magnetic resonance spectroscopy (1H-MRS).

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-60yo and generally healthy
2. BMI ≥ 25 kg/m2
3. Radiographic or histologic diagnosis of NAFLD / NASH
4. Insulin-like growth factor-1 (IGF-1) level <3rd quartile of normal for age

Exclusion Criteria:

1. Contraindications to MRI imaging
2. Diabetes mellitus or use of diabetes medications
3. History of cancer, significant renal disease, decompensated or unstable cardiovascular disease
4. Cirrhosis or known liver disease other than NAFLD
5. Pregnancy or breastfeeding
6. Known pituitary or hypothalamic disease affecting the growth hormone axis
7. Chronic use of drugs causing hepatic steatosis in the past 12 months (chronic oral steroids, methotrexate, tamoxifen)
8. Treatment with medications that may interact with LUM-201 (ibutamoren mesylate)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura E. Dichtel, MD, MHS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label Treatment
Started | 12
Completed | 7
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Baseline Liver Fat (Percent liver fat by 1H-MRS) [Mean (Standard Deviation); unit: percent liver fat] | 18.5 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Intrahepatic Lipid Content (IHL, Percent Liver Fat)
Description: Change in intrahepatic lipid content (6-month percent liver fat minus baseline percent liver fat) as measured by proton magnetic resonance spectroscopy (1H-MRS). Outcome is presented as change in percent liver fat.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: absolute change in percentage liver fat
Groups:
- Open-label Treatment With Ibutamoren: Open-label study of oral LUM-201 (ibutamoren mesylate) 25 mg daily in otherwise healthy adults with BMI ≥25 kg/m2 and NAFLD.
Arm/Group | Open-label Treatment With Ibutamoren
Number analyzed (Participants) | 7
absolute change in percentage liver fat | 3.9 (6.7)
Statistical Analysis 1: Comparison: Open-label Treatment With Ibutamoren; Subjects treated with open-label ibutamoren (n=7) were compared to historical placebo control subjects studied under identical inclusion criteria and procedures (n=10). The hypothesis is that open-label ibutamoren treatment would lead to a significant decrease in intrahepatic lipid content (IHL) as assessed by proton magnetic resonance spectroscopy (1H-MRS, absolute %IHL); Test type: Other; p = 0.4, t-test, 2 sided — Change in IHL over 6-months in absolute % IHL: Ibutamoren open-label 3.9 ± 6.7% versus historical placebo group 6.6 ± 6.1%, p=0.4

2. Secondary Outcome: Hepatic Inflammation and Fibrosis by LiverMultiScan Corrected T1 (cT1) Score
Description: Change in hepatic inflammation and fibrosis by LiverMultiScan cT1 (6-month cT1 score minus baseline cT1 score). Outcome is presented as change in cT1 score (ms). Higher values indicate more severe combined inflammation and fibrosis (normal range 633-794 ms).
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Open-label Treatment With Ibutamoren
Number analyzed (Participants) | 7
ms | 39 (44)
Statistical Analysis 1: Comparison: Open-label Treatment With Ibutamoren; Subjects treated with open-label ibutamoren (n=7) were compared to historical placebo control subjects studied under identical inclusion criteria and procedures (n=10). The hypothesis is that open-label ibutamoren treatment would lead to a significant decrease in hepatic inflammation and fibrosis as assessed by LiverMultiScan corrected T1 (cT1) score. There was no power calculation for this small pilot study; Test type: Other; p = 0.9, t-test, 2 sided — Change in cT1 over 6-months (ms): Ibutamoren open-label 39 ± 44 ms versus historical placebo group 44 ± 31 ms, p=0.9

3. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: Change in ALT (6-month ALT minus baseline ALT). Outcome is presented as change in ALT (U/L).
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Open-label Treatment With Ibutamoren
Number analyzed (Participants) | 7
U/L | 8 (18)
Statistical Analysis 1: Comparison: Open-label Treatment With Ibutamoren; Subjects treated with open-label ibutamoren (n=7) were compared to historical placebo control subjects studied under identical inclusion criteria and procedures (n=10). The hypothesis is that open-label ibutamoren treatment would lead to a significant decrease in alanine aminotransferase (ALT). There was no power calculation for this small pilot study; Test type: Other; p = 0.6, t-test, 2 sided — Change in ALT over 6-months (U/L): Ibutamoren open-label 8 ± 18 U/L versus historical placebo group 4 ± 8 U/L, p=0.6

ADVERSE EVENTS:
Time Frame: Adverse events were followed for each patient starting at the time of the screening period (minimum 0.5 months, maximum 3 months), during the six-month treatment phase (6 months), and for one month after the subject's last study visit. This represents a total time frame for adverse event assessment of approximately 7.5 months to 10 months.
Description: Adverse events are defined as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with drug exposure, whether or not considered related to drug exposure. Adverse events were assessed through regular investigator assessment at all study visits and at other points of patient contact between visits.
Arm/Group | Open-label Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Treatment (N=12)
Blurry vision (Eye disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Increased gas/bloating (Gastrointestinal disorders) | 2
Epigastric pain/GERD (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Night sweats (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ear infection (Ear and labyrinth disorders) | 1
Increased appetite (General disorders) | 7
Increased thirst/urination (General disorders) | 2
Upper respiratory infection (Infections and infestations) | 4 — 3 COVID+, 1 COVID negative
Brain fog (General disorders) | 1
Hyperglycemia (Endocrine disorders) | 4
Headaches (General disorders) | 2
Swelling of extremity (General disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 3
Weight gain (>5%) (Metabolism and nutrition disorders) | 1
Insomnia (General disorders) | 1
Nocturia (General disorders) | 1
Soreness at site of vaccine (General disorders) | 1
Vulvodynia (Reproductive system and breast disorders) | 1
Chest tightness/anxiety (General disorders) | 1
Congestion/cough (General disorders) | 1
Hypertension (General disorders) | 2
Groin/flank pain with kidney stone (Renal and urinary disorders) | 1
HPV+ on PAP (Infections and infestations) | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT05364684/Prot_SAP_000.pdf